CLINICAL TRIAL: NCT06721546
Title: The Effect of Healthy Nutrition and Functional Foods Education Based on the Health Promotion Model for Individuals With Type 2 Diabetes on Healthy Lifestyle Behaviors and Self-Efficacy in Diabetes: Randomized Controlled Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Oznur Gungor, nursing, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NecmettinEU/GÜNGÖR_001
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: type 2 diabetes, functional food, diabetes management, healthy eating
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Methods

STUDY DESIGN:
Intervention Model Description: This study aims to examine the effects of nursing interventions, including group training, reminder messages, and telephone counseling, based on a health promotion model, on healthy lifestyle behaviors related to the daily use of functional foods and diabetes self-efficacy among individuals aged 30-64 with Type 2 diabetes. The interventions were implemented through a researcher-prepared healthy nutrition and functional foods education booklet. The study employs a randomized pre-test-post-test controlled experimental design.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Other): The intervention group was provided with group education on healthy nutrition and functional foods based on the health promotion model, the provision of booklets, sending reminder messages and nursing interventions aimed at increasing motivation by providing telephone counseling. The intervention group was given an appointment for Tuesday-Thursday of the week for training at KEAH via telephone. After the training given to the intervention group, 2 reminder messages were given at two-week intervals and 3 telephone consultations were given, including the post-test application. 12 weeks after the training developed and applied according to the health promotion model given to the intervention group, post-test data were collected in both groups. In the post-test, the "Eating Habits and Functional Foods Information Form, Functional Food Consumption Form, Self-Efficacy Scale for Diabetes Management and Healthy Lifestyle Behaviors II" were applied as measurement tools.
  Interventions: Other: Nursing interventions; Other: reminder messages; Other: Telephone counseling
- control (No Intervention): In this group, type 2 diabetics were given pre-tests and post-tests (Functional Food Consumption Form, Diabetes Self-Efficacy Scale, Healthy Lifestyle Behaviors II Scale) during the pre-randomization phase during the familiarization phase between October 1 and October 30, 2024 during weekday daytime hours. No intervention was made to the control group. After the study was completed, the participants in the control group were given the right to be informed from an ethical perspective and a day was set for them to come to the hospital for 'healthy nutrition and functional food education' and education was started. The education is also provided in the booklet after the training.

INTERVENTIONS:
Other: Nursing interventions — The data collection process took place between March and June 2024. The implementation process took place between July 9 and October 24, 2024. In this process, education, reminder messages and telephone counseling for individuals with type 2 diabetes continued for 12 weeks.
  Introduction and Preliminary Preparation: Before randomization, both oral and written informed consent form and pretest forms (Personal Information Form, Nutrition Habits, Functional Foods Information Form, Functional Foods Consumption Form, Diabetes Self-Efficacy Scale, Healthy Lifestyle Behaviors II Scale Application) were administered by the researcher to individuals with type 2 diabetes who agreed to participate in the study between March and June 2024. After reaching the sample size (n=86), randomization was performed. Appointments were made for the intervention group for training at KEAH via telephone on Tuesday-Thursday of the week in groups.
  Arms: intervention
Other: reminder messages — Reminder messages: Address and telephone numbers of individuals with Type 2 diabetes in the intervention group were obtained after obtaining their informed consent at the first meeting. After the group training, the messages were sent to the groups (groups A, B, C and D) on Tuesdays and Thursdays during daylight hours every week on the 2nd (July 23-August 15) and 6th (August 20-September 12) weeks. The message was a reminder to the participants about healthy nutrition and consumption of functional foods.
  Arms: intervention
Other: Telephone counseling — Telephone counseling: After the group trainings applied to the intervention group, in the 4th (August 6-August 29) and 8th (September 3-September 26) weeks of each week on Tuesdays and Thursdays during daylight hours, individuals with diabetes mellitus were questioned about 'the obstacles they encounter during healthy eating and functional food consumption and whether they have the belief that they can overcome these obstacles and whether there is a change in their healthy eating and functional food consumption behaviors'. Reinforcement was made with reminder questions. In this process, the importance of functional food consumption was emphasized. The first telephone interview with 43 individuals with type 2 diabetes lasted 575 minutes in total and the second telephone interview lasted 495 minutes in total.
  Arms: intervention

SUMMARY:
Non-communicable diseases (NCDs) are defined by the World Health Organization (WHO) as "slowly progressing and long-lasting diseases, health problems that require continuous care due to the combination of genetic, physiological, environmental, and behavioral factors." (WHO 2023). One of these health issues, Diabetes Mellitus (DM), is one of the chronic and universal health problems affecting many people worldwide (Ministry of Health 2021). When diabetes is not controlled, many acute or chronic complications arise that significantly affect both the individual and society (Üstündağ and Dayapoğlu, 2021). As a result of the complications caused by diabetes, various organ and function losses occur in the individual. As a result, the individual's lifespan and quality of life are negatively affected, and social and economic losses that impact the entire society also occur. (Olgun ve ark. 2017). Therefore, healthy lifestyle behaviors influence minimizing the risk of diabetes and controlling the diabetes that has developed. These include healthy eating, regular medication use, regular exercise, weight maintenance, stress management, quitting smoking/alcohol, and patient education. Coordinating all of these ensures successful diabetes management (Üren and Karabulutlu 2018). Functional foods encompass certain minerals, fatty acids, dietary fibers (such as vegetables, fruits, whole grains, and legumes), antioxidants, or prebiotics that contain biologically active extracts and have beneficial effects on life. (Granato ve ark 2020). For example, foods that contain bioactive substances such as dietary fiber, polyphenols, saponins, and peptides, and have a low glycemic index, help diabetic patients in regulating their blood sugar levels. (Kazeem & Davies, 2016). Under the guise of nutrition education, natural functional foods that balance blood sugar in our daily lives can create awareness among individuals with type 2 diabetes, making diabetes management easier alongside medication treatment. To create a healthy society, ensuring that individuals and communities use healthy nutrition and functional foods in accordance with nutritional principles, based on their economic situations, will benefit the national economy and also improve the quality of life for individuals. Education conducted using a nursing model can further facilitate the adaptation process to chronic diseases. This study aims to examine the effects of nursing interventions, including group training, reminder messages, and telephone counseling, based on a health promotion model, on healthy lifestyle behaviors related to the daily use of functional foods and diabetes self-efficacy among individuals aged 30-64 with Type 2 diabetes. The interventions were implemented through a researcher-prepared healthy nutrition and functional foods education booklet. The study employs a randomized pre-test-post-test controlled experimental design. Before the random assignments of the 86 individuals who met the sample selection criteria and agreed to participate in the study into intervention and control groups, the Informed Consent Form, Personal Information Form, General Information Form on Eating Habits and Functional Foods, Functional Foods Consumption Form, Diabetes Self-Efficacy Scale, and Healthy Lifestyle Behaviors II Scale Form were completed. At the end of the 12th week after each group's training, the final tests will be conducted by the researcher via phone interview for the intervention and control groups. In the final test, the individuals in the intervention and control groups will be administered the General Information Form on Functional Foods, the Functional Food Consumption Form, the Healthy Lifestyle Behavior Scale-II, and the Self-Efficacy Scale for Diabetes Management in Diabetic Patients.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged 30-64 years
* Those diagnosed with Type 2 Diabetes for at least 6 months
* Not diagnosed with psychiatric and neurological diseases diagnosed by a doctor,
* Having basic diabetes knowledge,
* At least primary school graduate
* Individuals who volunteered to participate in the research,
* Smartphone and internet access,

Exclusion Criteria:

* Those who do not meet the inclusion criteria,
* Those who have a condition that prevents them from receiving education (physical, mental, vision and hearing, etc.)
* Those who have previously received functional food education,
* Those who are pregnant,
* Those with cancer,
* Those with acute or chronic kidney disease,
* Those with known food allergies.

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Healthy Lifestyle Behavior Scale-II | before randomization, at the time 12 weeks after education
  H0a: There is no difference between the mean scores of the healthy lifestyle behaviors assessment scale.
  H1a: There is a difference between the mean scores of the healthy lifestyle behaviors assessment scale.
Self-Efficacy Scale for Diabetes Management in Diabetes Patients | before randomization, at the time 12 weeks after education
  H0b: There is no difference between the mean scores of the self-efficacy in diabetes scale evaluation scale.
  H1b: There is a difference between the mean scores of the evaluation scale of the self-efficacy scale in diabetes.

SECONDARY OUTCOMES:
functional foods consumption form | before randomization, at the time 12 weeks after education

CONTACTS AND LOCATIONS:
Locations (1):
- Karaman education and research hospital, Karaman, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.who.int/news-room/fact-sheets/detail/noncommunicable-diseases